CLINICAL TRIAL: NCT00849277
Title: An RCT in Nursing Homes: the Effect of a Probiotic Treatment With Lactobacillus Casei Shirota on Respiratory Morbidity After Influenza Vaccination of Elderly.
Brief Title: Study of the Effect of Probiotics on Respiratory Morbidity After Influenza Vaccination of Elderly in Nursing Homes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Van Puyenbroeck Karolien, University of Antwerp
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2414
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2009-02-23 (Estimated); Status verified 2009-02

CONDITIONS: Respiratory Tract Infections
Keywords: Respiratory Tract Infections; Influenza, Human; Probiotics
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Lactobacillus casei Shirota

SUMMARY:
The purpose of this study is to determine whether probiotic treatment improves the protection against respiratory infections after influenza vaccination in elderly living in nursing homes.

DETAILED DESCRIPTION:
Influenza virus is a member of the orthomyxovirus family and causes an acute viral disease of the respiratory tract. The illness is usually self-limiting. Hospitalization and deaths mainly occur in high-risk groups (elderly, chronically ill). Response to vaccination is subject to high levels of variability due to age, stress, nutritional stage, etc.

Lactic acid bacteria are naturally commensal bacteria in the small and large intestines. These bacteria protect the host against potential pathogens by competitive exclusion and also by the production of antibacterial agents known as bacteriocins. It has only been recently shown that another mechanism whereby probiotic bacteria may provide a health benefit is by modulating immune responses.

Lactobacillus casei strain Shirota (LcS) is widely consumed in fermented milk products. Several studies, in animals as wells as in humans, report on the immunomodulatory functions of LcS.

The aim of this multicentre, randomized, placebo controlled, double blind study (RCT) is to assess if probiotic treatment with Lactobacillus casei Shirota improves the protection against influenza(-like) infections after vaccination with trivalent influenza vaccine in elderly residing in nursing homes.

Trial endpoints:

1. Clinical outcome: difference in incidence in upper respiratory tract infections (influenza-like illness)
2. Serological outcome: difference in influenza vaccine specific serum IgG between probiotic and control treatment

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female volunteers of 65 years or older
* volunteers reside in residential homes
* volunteers must be willing to swallow Yakult/placebo 2x/day for 3 weeks prevaccination and 5 months follow-up
* participants must be able to comply with requirements of study (e.g. assessment of respiratory symptoms, Yakult/placebo administration)
* participants must read and sign written Informed Consent Form after the nature of the study has been fully explained

Exclusion Criteria:

elderly with:

* any medical or practical condition which make the volunteer not suitable for participating in this study at discretion of the investigator
* any current relevant infectious disease
* any current known disorder having negative repercussions on the volunteer's immune system, such as auto-immune diseases, COPD requiring oxigen, cancer, chronic inflammatory disease
* allergy to influenza vaccine, eggs, neomycin, amphotericin B, erythromycin, amantadine
* ongoing treatment with immunosuppressive drugs, chemotherapeutics or other antineoplastic medication
* current use of antibiotics or use 6 weeks prior to study entry
* use of any investigative drug (other drugs who are also under investigation) within 90 days prior to study entry
* with markedly abnormal results in any of the screening laboratory tests

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 737 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Clinical outcome: difference in incidence in upper respiratory tract infections (influenza-like illness) | during 5 months
Serological outcome: difference in influenza vaccine specific serum IgG between probiotic and control treatment | 4 weeks after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] Van Puyenbroeck K, Hens N, Coenen S, Michiels B, Beunckens C, Molenberghs G, Van Royen P, Verhoeven V. Efficacy of daily intake of Lactobacillus casei Shirota on respiratory symptoms and influenza vaccination immune response: a randomized, double-blind, placebo-controlled trial in healthy elderly nursing home residents. Am J Clin Nutr. 2012 May;95(5):1165-71. doi: 10.3945/ajcn.111.026831. Epub 2012 Mar 21. PMID 22440853